CLINICAL TRIAL: NCT00079781
Title: RNS® System Feasibility Clinical Investigation
Brief Title: RNS® System Feasibility Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroPace (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NP10003
Record Dates: First submitted 2004-03-12; First posted 2004-03-16 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Epilepsy
Keywords: Responsive Stimulation; Brain Stimulator; Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Group (Active Comparator): Group of subjects who have undergone RNS® System implantation who are randomized to receive RNS® System responsive stimulation (i.e. responsive stimulation enabled or turned ON) during the blinded Evaluation Period. Stimulation is enabled during the first month post-implant and may continue throughout the subject's participation in the study.
  Interventions: Procedure: RNS® System implantation; Device: RNS® System responsive stimulation
- Sham Group (Sham Comparator): Group of subjects that have undergone RNS® System implantation that are randomized to receive sham-stimulation (i.e. responsive stimulation disabled or turned OFF) during the blinded Evaluation Period. Stimulation is enabled after transition into the Follow-Up Period (5th month post-implant) and may continue for the remainder of the subject's participation in the study.
  Interventions: Procedure: RNS® System implantation
- Open Label Group (Other): Group of subjects who have undergone RNS® System implantation who were not randomized or blinded to therapy status during the Evaluation Period. Stimulation may have been enabled during the first month post-implant and may have continued throughout the subject's participation in the study.
  Interventions: Procedure: RNS® System implantation; Device: RNS® System responsive stimulation

INTERVENTIONS:
Procedure: RNS® System implantation — Using standard neurosurgical techniques the surgical team implants the RNS® System, which includes the RNS® Neurostimulator and intracranial NeuroPace® Leads. Up to 4 Leads (Cortical Strips and/or Depth Leads) are placed in or near the epileptogenic focus/foci. The Neurostimulator is placed in the skull and connected to up to 2 Leads. At first the Neurostimulator is programmed to record brain activity (electrographic patterns). The neurologist or neurosurgeon reviews the recorded electrographic patterns and identifies abnormal (epileptiform, or seizure-like) activity. The Neurostimulator is then programmed to detect the abnormal activity.
Device: RNS® System responsive stimulation — The RNS® System is programmed to provide responsive stimulation (stimulation is ON or enabled). Upon detecting electrographic patterns, previously identified by the neurologist or neurosurgeon as abnormal (epileptiform, or seizure-like) activity, the Neurostimulator provides brief pulses of electrical stimulation through the Leads to interrupt those patterns. The typical patient is treated with a cumulative total of 5 minutes of stimulation a day.
  Arms: Open Label Group; Treatment Group

SUMMARY:
The RNS® System is intended to treat patients with medically refractory (hard to treat) epilepsy. The RNS® System Feasibility study is designed to demonstrate safety and evidence of effectiveness of the RNS® System to support the commencement of a pivotal clinical investigation.

DETAILED DESCRIPTION:
NeuroPace, Inc. is sponsoring an investigational device feasibility study of the RNS® System, the first closed loop responsive brain stimulator designed to treat medically refractory epilepsy. The RNS® System Feasibility study is a multi-center investigation being conducted at 12 epilepsy centers through the United States. The first 4 subjects at each site are entered into an open label protocol, and subsequent subjects at that site are entered into a randomized, double-blinded, sham-stimulation controlled protocol. The study is designed to demonstrate safety and evidence of effectiveness of the RNS® System to support commencement of a pivotal clinical investigation.

The RNS® Neurostimulator (a pacemaker-like device) and NeuroPace® Leads (tiny wires with electrodes) are implanted in the head. The Neurostimulator is a battery powered, microprocessor controlled device that detects and stores records of electrographic patterns (such as epileptiform, or seizure-like, activity) from the Leads within the brain. When the device detects an electrographic pattern, it responds by sending electrical stimulation through the Leads to a small part of the patient's brain to interrupt the electrographic pattern. This type of treatment is called responsive stimulation, but it is not yet known if it will work for the treatment of epilepsy. Direct brain stimulation therapy has already received approval in the United States, Europe, Canada, and Australia for the treatment of Essential Tremor and Parkinson's disease. Direct brain stimulation is not approved for the treatment of epilepsy.

Subjects participating in the RNS® System Feasibility study are required to have successfully completed the non-significant risk Prospective Seizure Frequency (PSF) study, which gathers baseline(pre-implant) seizure frequency data. Subjects must also met the inclusion criteria, including localization of epileptogenic region(s), prior to enrolling in the study. Throughout the entire study, subjects or their caregivers must keep a seizure diary. Seizure frequency, seizure severity, and antiepileptic medications, as well as physical and emotional health will be monitored and recorded throughout the study. Antiepileptic medications should continue to remain stable until 5 months post-implant.

Following enrollment, and prior to RNS® System implant, subjects undergo a neuropsychological evaluation. During the implant procedure, the RNS® Neurostimulator is cranially implanted and connected to one or two NeuroPace® Leads implanted in the brain. The investigational team determines the placement of the Leads based on prior localization of the epileptogenic region, according to standard localization procedures.

The Evaluation Period begins once the subject is implanted with the RNS® System and continues through the 4th month. Detection of epileptiform activity is enabled for all subjects within the first post-operative month. Responsive stimulation is enabled and optimized for subjects enrolled in the open label protocol or randomized to the Treatment group. Subjects randomized to the Sham group undergo simulated stimulation programming in order to maintain the treatment blind. Randomized subjects will not know whether responsive stimulation is being delivered or not.

At the beginning of the 5th month, subjects transition into the Follow up Period during which all subjects may receive responsive stimulation and antiepileptic medications may be adjusted as medically required. Subjects will be followed for 2 years post-implant. Throughout study participation, both effectiveness and safety data will be monitored continuously, and reviewed and documented by the study investigator at study appointments scheduled every 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has simple partial seizures (motor or sensory) or complex partial seizures (with motor manifestations) with or without secondarily generalized seizures
2. Subject has seizures that are distinct, stereotypical events that can be reliably counted, in the opinion of the investigator, by the subject or caregiver
3. Subject has seizures that are severe enough to cause injuries or significantly impair functional ability in domains including employment, psychosocial, education and mobility
4. Subject failed treatment with a minimum of two antiseizure medications (used in appropriate doses) with adequate monitoring of compliance and the effects of treatment
5. Subject has remained on the same antiseizure medication(s) over the preceding three (3) months (independent of dose and other than acute, intermittent use of benzodiazepines)
6. Subject has a minimum of four (4) or more countable seizures every month over the last three (3) months, as reported from the NeuroPace sponsored Prospective Seizure Frequency Clinical Investigation
7. Subject is ≥ 18 years old and ≤ 65 years old
8. Subject has undergone diagnostic testing that has established the epileptiform activity onset region(s) as part of his/her standard care to determine candidacy for epilepsy surgery
9. Subject is male, or if female is using a reliable method of contraception (hormonal, barrier method, surgical or abstention), or is at least two years postmenopause
10. Subject or legal guardian is able to provide appropriate consent to participate
11. Subject can be reasonably expected to maintain a seizure diary alone or with the assistance of a competent individual
12. Subject is able to complete regular office visits and telephone appointments per the protocol requirements
13. Subject is willing to be implanted with the RNS® System as a treatment for his/her seizures
14. Subject is able to tolerate a neurosurgical procedure
15. Subject is considered a good candidate to be implanted with an RNS® System

Note: 1 month = 28 days

Exclusion Criteria:

1. Subject has been diagnosed with psychogenic or non-epileptic seizures in the preceding year
2. Subject has been diagnosed with primarily generalized seizures
3. Subject has experienced unprovoked status epilepticus in the preceding year
4. In the opinion of the investigator, the subject has a clinically significant or unstable medical condition or a progressive central nervous system disease
5. Subject has been diagnosed with active psychosis, severe depression or suicidal ideation in the preceding year
6. Subject is pregnant or planning on becoming pregnant in the next year
7. Subject is on the ketogenic diet
8. Subject was enrolled in a therapeutic investigational drug or device study in the preceding year
9. Subject has an implanted Vagus Nerve Stimulator (VNS)
10. Subject has had therapeutic surgery to treat epilepsy in the preceding year
11. Subject is implanted with an electronic medical device that delivers electrical energy to the head or body
12. Subject is on chronic anticoagulants or, in the opinion of the investigator, subject is an unsuitable candidate for cranial surgery for any other reason
13. Subject had a cranial neurosurgical procedure in the previous month
14. Subject requires repeat MRIs
15. Subject's seizure onset zone(s) is/are located below the level of the subthalamic nucleus or, in the opinion of the investigator, the necessary lead placement would present too high a risk

Note: Subjects with an inactive VNS could be enrolled so long as the VNS was explanted prior to or at the same time as the RNS® System implant. Subjects who had had epilepsy surgery (resective, corpus callosotomy or ablation) greater than one year ago were still eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-01; Primary Completion 2006-05 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goodman, MD, Principal Investigator — Columbia University / Columbia Presbyterian Medical Center; Gregory Barkley, MD, Principal Investigator — Henry Ford Hospital; Greg Bergey, MD, Principal Investigator — Johns Hopkins University; Bruce Fisch, MD, Principal Investigator — Louisiana State University Epilepsy Center of Excellence; Robert Wharen, MD, Principal Investigator — Mayo Clinic; Richard Marsh, MD, Principal Investigator — Mayo Clinic; Richard Zimmerman, MD, Principal Investigator — Mayo Clinic; Anthony Murro, MD, Principal Investigator — Augusta University; Donna Bergen, MD, Principal Investigator — Rush University Medical Center / Epilepsy Center; Michael Smith, MD, Principal Investigator — Rush University Medical Center / Epilepsy Center; Ryder Gwinn, MD, Principal Investigator — Swedish Medical Center; Douglas Labar, MD, Principal Investigator — Weill Medical College of Cornell University; Robert Duckrow, MD, Principal Investigator — Yale University
Locations (12):
- United States (12):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center / Epilepsy Center, Chicago, Illinois
  - Louisiana State University Epilepsy Center of Excellence, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University / Columbia Presbyterian Medical Center, New York, New York
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Result] Barkley GL, Smith B, Bergey G, Worrell G, Chabolla D, Drazkowski J, Labar D, Duckrow R, Murro A, Smith M, Gwinn R, Fisch B, Hirsch L, and Morrell M. Safety and Preliminary Efficacy of the RNS Responsive Neurostimulator for the Treatment of Intractable Epilepsy in Adults. Epilepsia 2006; 47(S4):5.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Level 4 epilepsy centers, as categorized by the National Association of Epilepsy Centers (NAEC), through the United States.
Pre-assignment Details: In order to undergo initial implant, subjects were required to have successfully completed the non-significant risk Prospective Seizure Frequency (PSF) study, which gathered baseline characteristics and data including (pre-implant) seizure frequency. Subjects were required to maintain a minimum seizure frequency and remain on the same AED regimen.
Groups:
- Open Label Group: Group of subjects who underwent RNS® System implantation who were not randomized or blinded to therapy status during the Evaluation Period. Stimulation may have been enabled during the first month post-implant and may have continued throughout the subject's participation in the study.
- Treatment Group: Group of subjects who underwent RNS® System implantation who were randomized to receive RNS® System responsive stimulation (i.e. responsive stimulation enabled or turned ON) during the blinded Evaluation Period. Stimulation was enabled during the first month post-implant and may have continued throughout the subject's participation in the study.
- Sham Group: Group of subjects who underwent RNS® System implantation who were randomized to receive sham-stimulation (i.e. responsive stimulation disabled or turned OFF) during the blinded Evaluation Period. Stimulation may have been enabled after transition into the Follow-Up Period (5th month post-implant) and may have continued for the remainder of the subject's participation in the study.
Period: Pre-implant Period
Arm/Group | Open Label Group | Treatment Group | Sham Group
Started | 45 (Subjects were not assigned to a group until after initial implant.) | 10 (Subjects were not assigned to a group until after initial implant.) | 15 (Subjects were not assigned to a group until after initial implant.)
Completed | 42 (Subjects were not assigned to a group until after initial implant.) | 9 (Subjects were not assigned to a group until after initial implant.) | 14 (Subjects were not assigned to a group until after initial implant.)
Not Completed | 3 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Did not meet I/E criteria | 1 | 1 | 1
Period: Evaluation Period
Arm/Group | Open Label Group | Treatment Group | Sham Group
Started | 42 | 9 | 14
Completed | 42 | 9 | 14
Not Completed | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Open Label Group | Treatment Group | Sham Group
Started | 42 | 9 | 14
Completed | 38 | 9 | 12
Not Completed | 4 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Date of birth was not provided for 5 subjects (4 in the Open Label Group and 1 in the Treatment Group), therefore baseline characteristics calculations requiring age/DOB were derived using an N = 60.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label Group | Treatment Group | Sham Group | Total
Number analyzed (Participants) | 42 | 9 | 14 | 65
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 38 | 7 | 13 | 58
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (9.5) | 27.5 (7.6) | 36.2 (12.7) | 31.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 6 | 7 | 34
  Male | 21 | 3 | 7 | 31
Region of Enrollment [Number; unit: participants]
  United States | 42 | 9 | 14 | 65
Duration of epilepsy [Mean (Standard Deviation); unit: years] | 17.6 (10.4) | 17.4 (8.9) | 17.1 (10.3) | 17.5 (10.1)
Number of antiepileptic drugs (AEDs) used over lifetime [Mean (Standard Deviation); unit: AEDs] | 8.0 (2.6) | 7.3 (2.4) | 6.6 (2.7) | 7.6 (2.6)
Seizure onset location [Number; unit: participants]
  Mesial temporal lobe ONLY | 8 | 2 | 6 | 16
  Other | 34 | 7 | 8 | 49
Number of seizure foci [Number; unit: participants]
  Bifocal | 15 | 5 | 6 | 26
  Unifocal | 27 | 4 | 8 | 39
Prior intracranial monitoring for seizure localization [Number; unit: participants]
  Prior intracranial monitoring | 32 | 8 | 13 | 53
  NO prior intracranial monitoring | 10 | 1 | 1 | 12
Prior therapeutic surgery for epilepsy [Number; unit: participants]
  Prior therapeutic surgery for epilepsy | 18 | 2 | 4 | 24
  NO prior therapeutic surgery for epilepsy | 24 | 7 | 10 | 41
Prior vagal nerve stimulator (VNS) [Number; unit: participants]
  Yes | 16 | 0 | 2 | 18
  No | 26 | 9 | 12 | 47
Anatomical brain abnormality (by neuroimaging) [Number; unit: participants]
  Yes | 18 | 6 | 7 | 31
  No | 24 | 3 | 7 | 34

OUTCOME MEASURES:

1. Primary Outcome: Acute SAE Rate
Description: RNS® System Acute SAE Rate = the percentage of subjects having a serious adverse event (SAE) for the surgical implant procedure and the following month (28 days), whether reported as device-related or not.
  This outcome measure is met when the upper limit of the one-sided 95% confidence interval of the observed RNS® System Acute SAE Rate does not exceed the upper limit of the one-sided 95% confidence interval of the literature-based acute SAE rate associated with the implantation of intracranial electrodes for localization procedures and epilepsy surgery combined as documented in the literature (rate = 19%; upper CI = 28%). The comparator was calculated based upon the literature, therefore the number of participants analyzed is unknown/not applicable.
  The primary safety outcome measure was met.
Time Frame: Initial implant through 1 month post-implant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: Open Label Group, Treatment Group, and Sham Group combined.
Arm/Group | All Participants
Number analyzed (Participants) | 65
percentage of participants | 6.2 [2.4 to 14.8]

2. Primary Outcome: Short-term Chronic SAE Rate
Description: The RNS® System Short-term Chronic SAE rate = the percentage of implanted subjects having a serious adverse event (SAE) for the surgical implant procedure and the following 3 months (84 days), whether reported as device-related or not.
  This outcome measure is met when the upper limit of the one-sided 95% confidence interval of the observed RNS® System Short-term Chronic SAE Rate does not exceed the upper limit of the one-sided 95% confidence interval of the historical short-term chronic SAE rate for deep brain stimulation for movement disorders from the published literature (rate = 36%; upper CI = 46%). The comparator was calculated based upon the literature, therefore the number of participants analyzed is unknown/not applicable.
  The primary safety outcome measure was met.
Time Frame: Initial implant through 3 months post-implant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 65
percentage of participants | 9.2 [4.3 to 18.7]

3. Primary Outcome: Responder Rate
Description: Percentage of subjects with a 50% or greater reduction in mean seizure frequency during the post-implant Evaluation Period (4 months or 112 days) compared to pre-implant baseline (collected during the Prospective Seizure Frequency study). The primary effectiveness endpoint would be met with an observed responder rate of 13% or more.
  The effectiveness endpoint was only calculated for the Treatment Population. The endpoint was used to support a Pivotal Study, not to demonstrate efficacy when compared to a control/sham group.
  The primary effectiveness endpoint was met.
Time Frame: Pre-implant baseline through 4 months post-implant
Measure: Number; unit: Percent of participants
Groups:
- Treatment Population: Open Label Group and Treatment Group combined.
Arm/Group | Treatment Population
Number analyzed (Participants) | 51
Percent of participants | 24

ADVERSE EVENTS:
Time Frame: Initial implant through 2 years post-implant
Description: SAE = a positive or negative change in subject's physical/mental health as experienced by subject or observed by physician, during any part of the study, that resulted in:
  * significant risks/consequences to patient's acute or long-term health
  * serious injury or death
  * hospitalization or invasive medical intervention required to alleviate event
Groups:
- Sham Group: Group of subjects who underwent RNS® System implantation who were randomized to receive sham-stimulation (i.e. responsive stimulation disabled or turned OFF) during the blinded Evaluation Period). Stimulation may have been enabled after transition into the Follow-Up Period (5th month post-implant) and may have continued for the remainder of the subject's participation in the study.
Arm/Group | Treatment Population | Sham Group
Serious Adverse Events (participants affected / at risk) | 22/51 | 7/14
Other Adverse Events (participants affected / at risk) | 48/51 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Population (N=51) | Sham Group (N=14)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Biopsy lung (Investigations) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Complex partial seizures increased (Nervous system disorders) | 3 (3) | 0 (0)
Confusional state (Nervous system disorders) | 1 (1) | 0 (0)
Contusion (due to seizure) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Device lead damage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
EEG monitoring (Investigations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Implant site erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (due to seizure) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Live birth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 3 (3) | 1 (1)
Nonconvulsive status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postictal paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Premature battery depletion (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Psychiatric evaluation (Investigations) | 1 (1) | 0 (0)
Simple partial seizures increased (motor) (Nervous system disorders) | 1 (5) | 2 (3)
Skin laceration (due to seizure) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tonic-clonic seizures (Nervous system disorders) | 1 (1) | 0 (0)
Tonic-clonic seizures exacerbated (Nervous system disorders) | 1 (1) | 0 (0)
Tonic-clonic seizures increased (Nervous system disorders) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Population (N=51) | Sham Group (N=14)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Adverse drug reaction (General disorders) | 6 (7) | 0 (0)
Affect lability (Psychiatric disorders) | 2 (4) | 1 (1)
Agitation (Psychiatric disorders) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2)
Back injury (due to seizure) (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0)
Bradyphrenia (Nervous system disorders) | 3 (3) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Complex partial seizures (Nervous system disorders) | 3 (5) | 2 (2)
Complex partial seizures exacerbated (Nervous system disorders) | 1 (1) | 1 (1)
Complex partial seizures increased (Nervous system disorders) | 13 (19) | 6 (6)
Concussion (due to seizure) (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Confusional state (Nervous system disorders) | 3 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Contusion (due to seizure) (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Depression (Psychiatric disorders) | 8 (9) | 2 (2)
Depression suicidal (Psychiatric disorders) | 1 (1) | 2 (2)
Device interaction (General disorders) | 6 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 1 (2)
Diplopia (Eye disorders) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 3 (4) | 1 (1)
Dysaesthesia (Nervous system disorders) | 7 (7) | 1 (1)
Dysarthria (Nervous system disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 2 (2) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 1 (1)
Eyelid ptosis (Nervous system disorders) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (4)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hand fracture (due to seizure) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (due to seizure) (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 14 (22) | 5 (9)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 5 (5) | 1 (1)
Implant site discharge (General disorders) | 3 (4) | 0 (0)
Implant site pain (General disorders) | 10 (11) | 5 (5)
Implant site paraesthesia (General disorders) | 4 (4) | 1 (1)
Implant site swelling (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Influenza (Infections and infestations) | 5 (9) | 3 (7)
Ingrown hair (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 5 (6) | 4 (5)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (due to seizure) (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Libido decreased (Psychiatric disorders) | 5 (5) | 0 (0)
Memory impairment (Nervous system disorders) | 5 (5) | 3 (5)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Multiple injuries (due to seizure) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (21) | 3 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Night sweats (General disorders) | 2 (2) | 0 (0)
Nystagmus (Nervous system disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (4) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Photophobia (Nervous system disorders) | 1 (1) | 1 (1)
Photopsia (Nervous system disorders) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Post-traumatic headache (Nervous system disorders) | 2 (2) | 0 (0)
Postictal headache (Nervous system disorders) | 0 (0) | 2 (2)
Postoperative fever (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 24 (24) | 8 (8)
Procedural nausea (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 6 (8) | 0 (0)
Simple partial seizures (motor) (Nervous system disorders) | 5 (7) | 1 (4)
Simple partial seizures (sensory) (Nervous system disorders) | 3 (3) | 1 (1)
Simple partial seizures increased (motor) (Nervous system disorders) | 1 (1) | 2 (3)
Simple partial seizures increased (sensory) (Nervous system disorders) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Skin laceration (due to seizure) (Injury, poisoning and procedural complications) | 2 (9) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4) | 1 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 12 (17) | 7 (9)
Tonic-clonic seizures (Nervous system disorders) | 1 (1) | 2 (2)
Tonic-clonic seizures exacerbated (Nervous system disorders) | 3 (4) | 0 (0)
Tonic-clonic seizures increased (Nervous system disorders) | 3 (3) | 4 (4)
Tooth infection (Infections and infestations) | 2 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 8 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 4 (5) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2)
Visual disturbance (Eye disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5) | 1 (2)
Weight increased (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each Investigator, Coordinator, and Institution agree to submit publications to the RNS® System Study Publication Committee for review prior to submission for publication (at least 30 days for manuscripts and at least 7 days for abstracts) to assure that publication does not compromise the scientific integrity of the study or contain confidential NeuroPace information. NeuroPace may require that presentation/publication be withheld for up to 60 days to allow for filing of a patent application.